CLINICAL TRIAL: NCT03114917
Title: A Psychological Intervention for Suicide Applied to Patents With Psychosis: the CARMS Trial (Cognitive Approaches to Combatting Suicidality)
Brief Title: Cognitive AppRoaches to coMbatting Suicidality
Acronym: CARMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Greater Manchester Mental Health NHS Foundation Trust (Other); Lancaster University (Other)
Responsible Party: Principal Investigator, Patricia Gooding, Senior Lecturer, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/161/25; 220 (Other: Greater Manchester Mental Health NHS Foundation Trust)
Record Dates: First submitted 2017-03-29; First posted 2017-04-14 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Psychosis; Suicide Prevention; Suicidality
Keywords: Suicide; Self-harm; Psychosis; Community; Suicide Prevention; CBT; CARMS; Randomised controlled trial
MeSH Terms: conditions — Psychotic Disorders; Suicide Prevention; Suicidal Ideation; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Randomised-controlled trial with a qualitative component.
Who Masked: Outcomes Assessor
Masking Description: All Research Assistants will be blinded to treatment allocation. The Research Assistants will be carrying out outcomes assessments at baseline, 6 month and 12 month.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARMS therapy + TAU (Experimental): Participants allocated to the CARMS therapy + TAU arm will receive their usual care and treatment from mental health services along with CARMS (Cognitive AppRoaches to coMbatting Suicidality) therapy. The CARMS therapy comprises of 24 sessions, each up to 50 minutes long over a 6 month period.
  Interventions: Other: Cognitive AppRoaches to coMbatting Suicidality (CARMS)
- TAU (No Intervention): Participants allocated to treatment as usual (TAU) will receive their usual care and treatment from mental health services.

INTERVENTIONS:
Other: Cognitive AppRoaches to coMbatting Suicidality (CARMS) — The investigators' psychological therapy is a recovery-focused, structured, time-limited, socio-cognitive intervention. It is based upon the investigators' recently developed treatment manual (Tarrier et al., 2013) and pilot RCTs in the community (Tarrier et al., 2014) and in prison (Tarrier et al., accepted). The intervention modifies negative appraisals of emotional regulation, social support, and interpersonal problem-solving. As a consequence, perceptions of defeat, entrapment, and hopelessness will be improved indirectly. In addition, perceptions of defeat, entrapment, and hopelessness will be worked on directly during the therapy.
  Arms: CARMS therapy + TAU

SUMMARY:
This is a randomised controlled trial which investigates the effectiveness of CARMS (Cognitive AppRoaches to coMbatting Suicidality) therapy in reducing suicidal thoughts and how well CARMS works in practice within the NHS. The trial will compare two groups of people with psychosis who are using NHS mental health services. One group will carry on with their usual treatment. The other group will be offered 24 weekly sessions of CARMS therapy, plus their usual treatment.

DETAILED DESCRIPTION:
Estimates show that around 6% of people with experiences of psychosis die by suicide. Many more think about it and attempt suicide. A meta-analysis by the investigators illustrated that psychological therapies are effective in reducing suicidal thoughts and acts in people with psychosis as long as those therapies target suicidal thoughts, intentions and plans, and not the reduction of symptoms of mental illnesses. Based on this work, we have designed a psychological cognitive "talking" therapy (called CARMS) to reduce suicidal thoughts in people with experiences of psychosis which targets the psychological processes thought to underpin the pathways to suicidal thoughts and behaviours. An increasing body of work shows that many people with psychosis experience social isolation, emotional dysregulation, and poor interpersonal problem-solving. These appraisals can then induce and intensify perceptions of being hopeless, trapped and defeated, which in turn leads to suicidal thoughts and acts. CARMS aims to help people find practical ways to change these sorts of perceptions. Two of the investigators' pilot randomised trials have demonstrated that CARMS is feasible and acceptable to people experiencing psychosis and may have the potential to be effective at reducing key suicide outcomes.

Hence, the investigators' next step is to test the efficacy of CARMS in the context of NHS mental health services and also to test whether the underlying psychological mechanisms on which CARMS is based are correct. The investigators will test CARMS using a medium sized randomised controlled trial (RCT), with two arms of CARMS plus treatment as usual versus just treatment as usual. The target sample size is 250, with approximately 125 randomised to each arm of the trial, and an assumption of up to 25% attrition. Hence, the overall recruitment target is up to 333. The investigators will use both quantitative and qualitative methods and analyses to assess CARMS.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of psychosis (i.e. F20 - F29)
* suicidal thoughts and/or acts in the past three months
* in contact with mental health services and under the care of a mental health services clinical team (i.e., community or inpatient mental health care teams) with a care coordinator
* aged 18 or over
* English-speaking (hence, not needing an interpreter)
* able to give informed consent as assessed by either a responsible clinician or by trial RAs following the British Psychological Society's guidelines on gaining informed consent (http://www.bps.org.uk/sites/default/files/documents/code_of_human_research_ethics.pdf)

Exclusion Criteria:

* dementia, or an organic brain disorder
* unable to complete assessments due to language barriers
* currently taking part in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Adult Suicide Ideation Questionnaire score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Suicidal ideation valid measure

SECONDARY OUTCOMES:
Change from Baseline Suicide Probability Scale score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Suicide risk valid measure
Change from Baseline Beck Scale for Suicidal ideation score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Assess an individual's thoughts, attitudes and intentions regarding suicide
Change from Baseline Frequency of suicidal thoughts, plans and acts at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Clinical interview to ascertain frequency of suicidal thoughts, plans and acts across six months
Change from Baseline Frequency of Suicide Attempts at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Frequency of suicide attempts will be collected from medical records

OTHER OUTCOMES:
Change from Baseline Difficulties in Emotional Regulation Scale score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  The questionnaire measures emotional dysregulation
Change from Baseline Social Problem-Solving Inventory score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  The questionnaire measures individual's social problem-solving skills
Change from Baseline Social Support Appraisals Scale score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  The questionnaire measures individual's appraisals of social support
Change from Baseline Beck Hopelessness Scale score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  The questionnaire measures three aspects of hopelessness: feelings about the future, loss of motivation, and expectations
Change from Baseline Defeat and Entrapment scale scores at 6 and 12 months | Baseline, 6 month and 12 month follow up
  The questionnaire measures how defeated and trapped individuals feel respectively
Change from Baseline Positive and Negative Syndrome Scale score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Clinical interview to assess symptom severity of individual's experiencing Schizophrenia
Change from Baseline Psychotic Symptoms Ratings Scale (PSYRATS) score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Clinical interview to assess symptoms of psychosis
Change from Baseline Personal and Social Performance Scale score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Clinical interview to assess personal and social functioning in individual's experiencing Schizophrenia
Change from Baseline Calgary Depression Scale score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Clinical interview to assess symptoms of depression in individual's experiencing Schizophrenia
Change from Baseline Frequency and Type of Substance Misuse as measured by the Timeline Follow Back at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Clinical interview to ascertain frequency and type of substance misuse over 3 months
Change from Baseline Drug use (self-reported) DAST score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Measure which identifies drug 'abuse'
Change from Baseline Alcohol use (self-reported) AUDIT score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Gold standard measure which identifies alcohol use
Change from Baseline Reasons for substance Use Scale - Alcohol and Drugs scores at 6 and 12 months | Baseline, 6 month and 12 month follow up
  Questionnaire measure which identifies individual's reasons for using alcohol and drugs respectively
Change from Baseline Sleep Condition Indicator score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  The questionnaire measures insomnia
Current medication for mental health problems as prescribed at baseline assessment time point | Baseline
  Information regarding which anti-psychotic medication, if the medication is atypical, and the dosage will be collected from medical records
Change from Baseline Working Alliance Inventory - short form score at 6 and 12 months | Baseline, 6 month and 12 month follow up
  The questionnaire measure the client-therapist therapeutic alliance from the participant's and the therapist's perspective
Change from Baseline EQ-5D score at 12 months | Baseline and 12 month follow up
  The questionnaire measures health outcomes
Change from Baseline Client Service Use Receipt Inventory at 12 months | Baseline and 12 month follow up
  The questionnaire measures use of services

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Gooding, Principal Investigator — University of Manchester; Gillian Haddock, Principal Investigator — University of Manchester
Locations (4):
- United Kingdom (4):
  - Pennine Care NHS Foundation Trust, Ashton-under-Lyne
  - Lancashire Care NHS Foundation Trust, Chorley
  - Greater Manchester Mental Health NHS Trust, Manchester
  - Northwest Boroughs Healthcare NHS Foundation Trust, Warrington

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are undecided at present.

REFERENCES:
- [Derived] Gooding P, Pratt D, Edwards D, Awenat Y, Drake RJ, Emsley R, Jones S, Kapur N, Lobban F, Peters S, Boardman B, Harris K, Huggett C, Haddock G. Underlying mechanisms and efficacy of a suicide-focused psychological intervention for psychosis, the Cognitive Approaches to Combatting Suicidality (CARMS): a multicentre, assessor-masked, randomised controlled trial in the UK. Lancet Psychiatry. 2025 Mar;12(3):177-188. doi: 10.1016/S2215-0366(24)00399-7. Epub 2025 Jan 16. PMID 39827886
- [Derived] Gooding P, Haddock G, Harris K, Asriah M, Awenat Y, Cook L, Drake RJ, Emsley R, Huggett C, Jones S, Lobban F, Marshall P, Pratt D, Peters S. The interplay between suicidal experiences, psychotic experiences and interpersonal relationships: a qualitative study. BMC Psychiatry. 2023 Nov 24;23(1):873. doi: 10.1186/s12888-023-05164-2. PMID 38001403
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Gooding PA, Pratt D, Awenat Y, Drake R, Elliott R, Emsley R, Huggett C, Jones S, Kapur N, Lobban F, Peters S, Haddock G. A psychological intervention for suicide applied to non-affective psychosis: the CARMS (Cognitive AppRoaches to coMbatting Suicidality) randomised controlled trial protocol. BMC Psychiatry. 2020 Jun 16;20(1):306. doi: 10.1186/s12888-020-02697-8. PMID 32546129